CLINICAL TRIAL: NCT00993473
Title: A 24-week, Randomized, Open-label, Parallel Group Multinational Comparison of Lantus® (Insulin Glargine) Given in the Morning as Once-a-day Basal Insulin Versus Neutral Protamine Hagedorn (NPH) Insulin, in Children With Type 1 Diabetes Mellitus Aged at Least 1 Year to Less Than 6 Years
Brief Title: 6-month Comparison of Morning Lantus Versus Neutral Protamine Hagedorn Insulin in Young Children With Type 1 Diabetes
Acronym: PRESCHOOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11202; 2009-011231-12 (EudraCT Number)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2012-06-22 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lantus (insulin glargine) (Experimental): Lantus given as basal insulin once a day in the morning by subcutaneous injection
  Interventions: Drug: Insulin glargine (HOE901); Drug: Insulin lispro
- NPH insulin (Active Comparator): Neutral Protamine Hagedorn (NPH) human insulin given as basal insulin either once or twice per day generally in the morning and /or at bedtime by subcutaneous injection
  Interventions: Drug: Neutral Protamine Hagedorn (NPH) insulin; Drug: Insulin lispro

INTERVENTIONS:
Drug: Insulin glargine (HOE901) — 100 U/mL commercial solution for injection available as both disposable pen devices Solostar® each containing 300 U and as 10 mL vials each containing 1000 U
  Dose: titrated to achieve the following glycemic targets without hypoglycemia:
  * Fasting blood glucose (BG) between 90 and 145 mg/dL (5.0 to 8.0 mmol/L), inclusive,
  * Bedtime BG between 120 and 180 mg/dL (6.7 to10.0 mmol/L), inclusive,
  * Nocturnal BG between 80 and 162 mg/dL (4.4 to 9.0 mmol/L), inclusive; and
  * HbA1c <7.5%.
  Other Names: Lantus®
  Arms: Lantus (insulin glargine)
Drug: Neutral Protamine Hagedorn (NPH) insulin — NPH insulin 100 U/mL commercial (Huminsulin Basal) solution for injection available as both disposable pen devices (Huminsulin Basal Pen) each containing 300 U and as 10 mL vials each containing 1000 U
  Dose: titrated to achieve glycemic targets as described above for insulin glargine
  Arms: NPH insulin
Drug: Insulin lispro — Insulin lispro used as the principal bolus insulin; regular human insulin permitted. Administration: multiple injection before meals and/or at bedtime at the discretion of the Investigator.
  Other Names: Humalog®

SUMMARY:
The primary study objective was to compare the rate of "all hypoglycemia" (composite outcome of the following hypoglycemia events: symptomatic hypoglycemia episodes, low continuous glucose monitoring system (CGMS) excursions confirmed by fingerstick blood glucose (FSBG), low FSBG readings performed at other times) between children treated with Lantus (insulin glargine) and Neutral Protamine Hagedorn (NPH) insulin.

Secondary objectives were to compare insulin glargine and NPH in terms of:

* rates of specific types of hypoglycemia: symptomatic, severe, nocturnal, nocturnal symptomatic, and severe nocturnal symptomatic hypoglycemia
* HbA1c change from baseline to end-of-treatment, and HbA1c at end-of-treatment
* percentage of patients reaching HbA1c less than 7.5% (target value) at end of treatment
* average blood glucose over whole trial and at end of trial, as estimated by continuous glucose monitoring (CGM), and blood glucose variability

DETAILED DESCRIPTION:
Screening phase: 2 to 4 weeks

Treatment phase: 24 weeks

At randomization, patients were stratified with respect to their baseline HbA1c level (<8.5% or ≥8.5%) and hypoglycemic event rate (number of CGMS hypoglycemic excursions <0.5 or ≥0.5 events per 24 hours). Following randomization, trial basal insulin was initiated and up-titrated within the first 12 weeks to reach a stable dose.

Follow-up phase: 2 weeks

All Phases: 28 to 30 weeks

ELIGIBILITY:
Inclusion criteria:

* Pediatric patients with type 1 diabetes mellitus aged at least one year to less than 6 years at screening, for whom signed written informed consent has been obtained from parent or legal guardian to participate in the study

Exclusion criteria:

* Diagnosis of type 1 diabetes for less than one year
* HbA1c at screening >12% or <6%
* Diabetes other than type 1 diabetes
* Parents and patients not willing to undergo all study assessments and treatments, including home blood glucose monitoring, Continuous Glucose Monitoring System (CGMS) sensor placement and maintenance both at the site and at home, multiple daily insulin injections, and visits, as dictated by the protocol (if a telephone is not available patients may undergo all visits in person)
* Patients and families for whom 6 days in total (not necessarily continuous) of useable CGMS data cannot be obtained (either by home sensor replacement, or by sensor replacement at the site at additional screening visits if needed) during the screening CGMS evaluations between Visit 2 and the randomization visit
* Patients treated with insulin pump therapy during the two months prior to screening
* History of primary seizure disorder
* History of severe hypoglycemic episode accompanied by seizure and/or coma, or diabetic ketoacidosis leading to hospitalization or to care in the emergency ward, in the 2 months prior to the screening visit
* Need for chronic treatment with acetaminophen (paracetamol)-containing medications
* Serum creatinine > 2.0mg/dL at screening
* Serum ALT or AST greater than 3x upper limit of normal for the patient's age and gender, at screening
* Hemoglobin < 10g/dL, or platelet count less than 100,000/cu mm, at screening
* Treatment with any pharmacologic anti-hyperglycemic oral agent for more than 3 months at any time
* Treatment with any non-insulin antihyperglycemic medication (eg, Symlin®) for the 3 months prior to screening
* Treatment with systemic glucocorticoids within the month prior to screening

Above information not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (61):
- United States (8):
  - Sanofi-Aventis Investigational Site Number 840006, Sacramento, California
  - Sanofi-Aventis Investigational Site Number 840014, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840005, Greenwood Village, Colorado
  - Sanofi-Aventis Investigational Site Number 840008, Baltimore, Maryland
  - Sanofi-Aventis Investigational Site Number 840007, Buffalo, New York
  - Sanofi-Aventis Investigational Site Number 840011, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840010, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840002, San Antonio, Texas
- Sanofi-Aventis Investigational Site Number 040001, Vienna, Austria
- Brazil (6):
  - Sanofi-Aventis Investigational Site Number 076001, Brasília
  - Sanofi-Aventis Investigational Site Number 076003, Curitiba
  - Sanofi-Aventis Investigational Site Number 076005, Fortaleza
  - Sanofi-Aventis Investigational Site Number 076004, Fortaleza
  - Sanofi-Aventis Investigational Site Number 076002, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076006, Rio de Janeiro
- Chile (4):
  - Sanofi-Aventis Investigational Site Number 152002, Santiago
  - Sanofi-Aventis Investigational Site Number 152003, Santiago
  - Sanofi-Aventis Investigational Site Number 152001, Santiago
  - Sanofi-Aventis Investigational Site Number 152004, Viña del Mar
- Czechia (3):
  - Sanofi-Aventis Investigational Site Number 203001, Olomouc
  - Sanofi-Aventis Investigational Site Number 203003, Pardubice
  - Sanofi-Aventis Investigational Site Number 203002, Ústí nad Labem
- Germany (2):
  - Sanofi-Aventis Investigational Site Number 276002, Düsseldorf
  - Sanofi-Aventis Investigational Site Number 276003, Münster
- Hungary (5):
  - Sanofi-Aventis Investigational Site Number 348004, Budapest
  - Sanofi-Aventis Investigational Site Number 348005, Budapest
  - Sanofi-Aventis Investigational Site Number 348003, Miskolc
  - Sanofi-Aventis Investigational Site Number 348002, Szeged
  - Sanofi-Aventis Investigational Site Number 348001, Szombathely
- India (5):
  - Sanofi-Aventis Investigational Site Number 356003, Bangalore
  - Sanofi-Aventis Investigational Site Number 356005, Bangalore
  - Sanofi-Aventis Investigational Site Number 356001, Bangalore
  - Sanofi-Aventis Investigational Site Number 356002, Indore
  - Sanofi-Aventis Investigational Site Number 356004, Karnāl
- Mexico (3):
  - Sanofi-Aventis Investigational Site Number 484002, Guadalajara
  - Sanofi-Aventis Investigational Site Number 484003, Monterrey
  - Sanofi-Aventis Investigational Site Number 484001, Puebla City
- Peru (3):
  - Sanofi-Aventis Investigational Site Number 604003, Lima
  - Sanofi-Aventis Investigational Site Number 604002, Lima
  - Sanofi-Aventis Investigational Site Number 604001, Lima
- Poland (2):
  - Sanofi-Aventis Investigational Site Number 616002, Gdansk
  - Sanofi-Aventis Investigational Site Number 616001, Warsaw
- Romania (4):
  - Sanofi-Aventis Investigational Site Number 642008, Bucharest
  - Sanofi-Aventis Investigational Site Number 642001, Cluj-Napoca
  - Sanofi-Aventis Investigational Site Number 642011, Constanța
  - Sanofi-Aventis Investigational Site Number 642006, Sibiu
- Russia (5):
  - Sanofi-Aventis Investigational Site Number 643001, Moscow
  - Sanofi-Aventis Investigational Site Number 643002, Moscow
  - Sanofi-Aventis Investigational Site Number 643003, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643004, Ufa
  - Sanofi-Aventis Investigational Site Number 643005, Yaroslavl
- South Africa (4):
  - Sanofi-Aventis Investigational Site Number 710004, Durban
  - Sanofi-Aventis Investigational Site Number 710002, Johannesburg
  - Sanofi-Aventis Investigational Site Number 710001, Observatory
  - Sanofi-Aventis Investigational Site Number 710003, Pretoria
- Spain (4):
  - Sanofi-Aventis Investigational Site Number 724003, Santiago de Compostela
  - Sanofi-Aventis Investigational Site Number 724001, Seville
  - Sanofi-Aventis Investigational Site Number 724005, Valencia
  - Sanofi-Aventis Investigational Site Number 724004, Zaragoza
- Turkey (Türkiye) (2):
  - Sanofi-Aventis Investigational Site Number 792001, Ankara
  - Sanofi-Aventis Investigational Site Number 792003, Istanbul

REFERENCES:
- [Derived] Danne T, Becker RH, Ping L, Philotheou A. Insulin glargine metabolite 21(A) -Gly-human insulin (M1) is the principal component circulating in the plasma of young children with type 1 diabetes: results from the PRESCHOOL study. Pediatr Diabetes. 2015 Jun;16(4):299-304. doi: 10.1111/pedi.12161. Epub 2014 Jul 9. PMID 25041275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 61 centers (72 were initiated) in 16 countries between October 15, 2009 and March 30, 2011.
Pre-assignment Details: A total of 165 patients were screened and 125 were randomized. Forty patients (24.2%) failed the screening selection process, mainly due to noncompliance with the study required Continuous Glucose Monitoring (CGM) performance and other procedures.
Groups:
- Lantus (Insulin Glargine): Lantus (insulin glargine) given as basal insulin once a day in the morning by subcutaneous injection.
  Dose: titrated to achieve glycemic targets as described in protocol section.
- NPH Insulin: Neutral Protamine Hagedorn (NPH) human insulin given as basal insulin either once or twice per day by subcutaneous injection.
  Dose: titrated to achieve glycemic targets as described in protocol section.
Period: Overall Study
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Started | 61 (61 patients randomized to Lantus but 62 patients treated with Lantus due to a dispensation's error) | 64 (64 patients randomized to NPH but only 63 patients treated with NPH due to a dispensation's error)
Completed | 57 | 54
Not Completed | 4 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Technical problem with CGM device | 0 | 1
Not completed — Family event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin | Total
Number analyzed (Participants) | 61 | 64 | 125
Age Continuous [Mean (Standard Deviation); unit: years] | 4.3 (0.9) | 4.1 (1.0) | 4.2 (1.0)
Age Continuous [Median (Full Range); unit: years] | 5.0 [2 to 5] | 4.0 [1 to 6] | 4.0 [1 to 6]
Age, Customized [Number; unit: participants]
  <= 3 years | 10 | 17 | 27
  > 3 years | 51 | 47 | 98
Sex/Gender, Customized [Number; unit: participants]
  Male | 32 | 30 | 62
  Female | 29 | 34 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 53 | 48 | 101
  Black | 2 | 2 | 4
  Asian/Oriental | 4 | 11 | 15
  Other | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 17 | 13 | 30
  Non Hispanic | 44 | 51 | 95
Duration of diabetes [Mean (Standard Deviation); unit: years] | 2.12 (1.16) | 2.12 (1.01) | 2.12 (1.08)
Duration of diabetes [Median (Full Range); unit: years] | 1.63 [1.0 to 5.3] | 2.05 [1.0 to 4.9] | 1.81 [1.0 to 5.3]
Treated by bolus insulin at baseline [Number; unit: participants]
  Yes | 54 | 58 | 112
  No | 7 | 6 | 13
Treated by basal insulin at baseline [Number; unit: participants]
  Yes | 58 | 57 | 115
  No | 3 | 7 | 10
Treated by mixed (bolus & basal) insulin at baseline [Number; unit: participants]
  Yes | 5 | 8 | 13
  No | 56 | 56 | 112
Number of daily basal insulin injections at baseline [Number; unit: participants]
  1 | 32 | 41 | 73
  2 | 21 | 15 | 36
  >=3 | 5 | 1 | 6
  Not treated with basal insulin at baseline | 3 | 7 | 10
Total daily dose of basal insulin injection at baseline [Number; unit: participants]
  Analyzed | 57 | 57 | 114
  Not treated by basal insulin or missing | 4 | 7 | 11
Total daily dose of basal insulin injection at baseline [Mean (Standard Deviation); unit: International Units] | 7.29 (4.11) | 7.61 (4.77) | 7.45 (4.43)
Total daily dose of basal insulin injection at baseline [Median (Full Range); unit: International Units] | 6.00 [2.0 to 24.0] | 6.00 [1.5 to 24.0] | 6.00 [1.5 to 24.0]
Total daily dose of bolus insulin injection at baseline [Number; unit: participants]
  Analyzed | 52 | 57 | 109
  Not treated by bolus insulin or missing | 9 | 7 | 16
Total daily dose of bolus insulin injection at baseline [Mean (Standard Deviation); unit: International Units] | 7.14 (3.64) | 7.98 (7.20) | 7.58 (5.77)
Total daily dose of bolus insulin injection at baseline [Median (Full Range); unit: International Units] | 7.75 [1.3 to 16.0] | 7.00 [0.8 to 45.0] | 7.00 [0.8 to 45.0]

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of "All Hypoglycemia" Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years (Events Per Patient-year)
Description: The rate of "all hypoglycemia" was calculated from "all hypoglycemia" episodes which occurred during the 24-week on-treatment period and consisted of: - symptomatic hypoglycemia episodes validated by the study investigator based on entries in patients' diaries, - low continuous glucose monitoring system (CGMS) excursions (interstitial glucose <70 mg/dL [3.9 mmol/L]) confirmed by fingerstick blood glucose (FSBG) <70 mg/dL, - low FSBG readings (values <70 mg/dL) performed at other times.
Time Frame: 6 months
Population: The efficacy population consisted of all randomized patients who received at least one dose of the study medication (modified intent-to-treat [mITT] population). For efficacy analyses, patients were analyzed in the treatment group allocated by the Interactive Voice Response System (IVRS) at randomization (as randomized).
Measure: Mean (Standard Deviation); unit: number of events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
number of events per patient-year | 192.75 (119.28) | 168.91 (101.04)
Statistical Analysis 1: Comparison: Lantus (Insulin Glargine) vs NPH Insulin; The sample size was calculated to ensure sufficient power so that the upper bound of the 2-sided 95% CI for the Lantus /NPH ratio would not exceed 1.15 based on an expected overall rate of "all hypoglycemia" of 80 events per patient-year of exposure to NPH insulin and to Lantus. It was planned to randomize at least 45 and up to approximately 60 patients in each of the 2 treatment groups so that at least 70 patients would complete the 24 weeks of treatment; Test type: Non-Inferiority or Equivalence — Noninferiority would be demonstrated if the upper bound of the 95% confidence interval (CI) for the ratio of the rate of "all hypoglycemia" in the Lantus group to the rate in the NPH group was <1.15. Superiority would be demonstrated if the upper bound of the 95% CI was <1. The margin for noninferiority corresponded to one-half of the 30% difference in hypoglycemia event rate considered as a clinically significant difference by American Diabetes Association 2005 Working Group on Hypoglycemia; Generalized Linear Model; A stepwise closed testing approach was used for the primary "all hypoglycemia" outcome analysis to assess noninferiority and superiority sequentially; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.97 to 1.44], Standard Error of Mean 0.12 — Risk ratio between treatment groups (Lantus/NPH) estimated by Generalized Linear Model with fixed effect terms for randomization strata and treatment

2. Secondary Outcome: Event Rate of Symptomatic Hypoglycemia (Individual Component of Primary Endpoint) Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years (Events Per Patient-year)
Description: Symptomatic hypoglycemia: any event with clinical symptoms considered to result from hypoglycemia, validated by the study investigator based on data from patient diaries.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
events per patient-year | 25.54 (37.25) | 33.02 (47.95)

3. Secondary Outcome: Event Rate of Severe Symptomatic Hypoglycemia Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years
Description: Severe symptomatic hypoglycemia: any event with clinical symptoms considered to result from a hypoglycemic episode for which the patients required the assistance of a third party (ie, other than the patient, or a parent/usual caregiver; eg, from emergency personnel), because the patients/parents could not treat the event with acute neurological impairment directly resulting from the hypoglycemic event. The occurrence of seizure, coma, unconsciousness, or the use of glucagon, were also to qualify a hypoglycemic episode as severe.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: number of events per patient-year
Units Other Than Participants: Episodes
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
Number analyzed (Episodes) | 4 | 2
number of events per patient-year | 0.14 (0.55) | 0.07 (0.38)

4. Secondary Outcome: Event Rate of Nocturnal Hypoglycemia Defined as the Total Number of "All Hypoglycemia" Episodes Divided by the Total Duration of the On-treatment Period in Years
Description: Nocturnal hypoglycemia: any event from the "all hypoglycemia" total that occurred between 23:00 and 07:00 hours.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: number of events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
number of events per patient-year | 33.50 (25.62) | 30.92 (24.97)

5. Secondary Outcome: Event Rate of Nocturnal Symptomatic Hypoglycemia Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years
Description: Nocturnal symptomatic hypoglycemia: any symptomatic hypoglycemic event that occurred between 23:00 and 07:00 hours.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: number of events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
number of events per patient-year | 2.38 (5.42) | 3.65 (6.75)

6. Secondary Outcome: Event Rate of Severe Nocturnal Hypoglycemia Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years
Description: Severe nocturnal symptomatic hypoglycemia: any severe symptomatic hypoglycemic event that occurred between 23:00 and 07:00 hours.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: number of events per patient-year
Units Other Than Participants: Episodes
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
Number analyzed (Episodes) | 1 | 0
number of events per patient-year | 0.04 (0.29) | 0.00 (0.00)

7. Secondary Outcome: Glycosylated Hemoglobin A1c (HbA1c): End of Treatment and Change From Baseline to End of Treatment
Time Frame: baseline, 6 months
Population: Same as for primary endpoint: mITT population. However post-baseline HbA1c values were missing for 9 patients: 2 patients in the Lantus group and 7 in the NPH group.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
percent HbA1c
  Baseline HbA1c | 8.023 (1.049) | 8.248 (1.429)
  End of treatment HbA1c (N = 59 & 57) | 8.071 (0.884) | 8.344 (1.161)
  Absolute change from baseline (N = 59 & 57) | 0.036 (0.979) | 0.000 (1.035)

8. Secondary Outcome: Glycosylated Hemoglobin A1c (HbA1c): End of Treatment and Change From Baseline to End of Treatment (ANCOVA Estimates)
Description: Assessed using an analysis of covariance (ANCOVA) model with treatment, and randomization strata (baseline number of CGM hypoglycemic excursions <0.5 events/24hours or ≥0.5 events/24 hours, and baseline HbA1c <8.5% or ≥8.5%) as fixed effects, and using the baseline value as covariate.
Time Frame: baseline, 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent HbA1c
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
percent HbA1c
  End of treatment HbA1c (ANCOVA) | 8.139 (0.1065) | 8.232 (0.1134)
  Absolute change from baseline HbA1c (ANCOVA) | -0.048 (0.1065) | 0.045 (0.1134)

9. Secondary Outcome: Percentage of Patients Reaching HbA1c Target of Less Than 7.5% at the End of Treatment Visit
Description: Percentage of patients reaching International Society for Pediatric and Adolescent Diabetes (ISPAD)-recommended goals of Glycosylated Hemoglobin A1c <7.5% at the end of treatment visit.
Time Frame: 6 months
Population: The population analyzed consisted of patients from the mITT population (as defined for primary outcome measure) with post-baseline HbA1c values. 2 patients from the Lantus group and 7 from the NPH group had no post-baseline HbA1c value.
Measure: Number; unit: percentage of participants
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 59 | 57
percentage of participants | 22.0 | 22.8

10. Secondary Outcome: Average Daily Blood Glucose (BG) Based on CGMS Values: End of Treatment and Change From Baseline to End of Treatment
Time Frame: baseline, 6 months
Population: Same as for primary endpoint: mITT population. However 1 patient in the NPH group did not have baseline CGM value and 2 other patients (1 in the Lantus group and 1 in the NPH group) did not have on-treatment CGM values.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
mmol/L
  Baseline daily BG (N= 61 & 63) | 11.263 (1.887) | 11.170 (1.986)
  End of treatment daily BG (N= 60 & 63) | 11.085 (2.077) | 11.712 (2.166)
  Absolute change from baseline (N= 60 & 62) | -0.218 (2.399) | 0.501 (1.906)

11. Other Pre Specified Outcome: Number of Patients With Different Types of Hypoglycemia Events
Description: Definitions of the different types of hypoglycemia events provided in the outcome measure description of the corresponding event rates.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Number; unit: participants
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
participants
  Patients with "All hypoglycemia" | 61 | 63
  Patients with symptomatic hypoglycemia | 40 | 44
  Patients with severe symptomatic hypoglycemia | 4 | 2
  Patients with nocturnal hypoglycemia | 59 | 60
  Patients with nocturnal symptomatic hypoglycemia | 17 | 28
  Patients with severe noct. sympto. hypoglycemia | 1 | 0
  Patients with "All confirmed low CGMS excursions" | 60 | 61
  Patients with "All confirmed low FSBG" | 61 | 63

12. Other Pre Specified Outcome: Percent of Blood Glucose (BG) Within the Range of 70 - 180 mg/dL (3.9-10 mmol/L)
Description: Calculated for each patient as the percent of all on-treatment CGMS values falling within the range of 70 - 180 mg/dL (3.9 - 10 mmol/L) inclusive.
Time Frame: 6 months
Population: The population analyzed consisted of patients from the mITT population (as defined for primary outcome measure) with on-treatment CGM values (1 patient from the Lantus group and 1 from the NPH group did not have on-treatment CGM).
Measure: Mean (Standard Deviation); unit: percent of CGMS values within the range
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 60 | 63
percent of CGMS values within the range | 41.667 (12.048) | 38.158 (10.908)

13. Other Pre Specified Outcome: Blood Glucose Variability Based on All On-treatment CGMS Values
Description: Calculated for any given patient as the standard deviation (SD) of all CGMS interstitial glucose values recorded over all CGMS placements.
Time Frame: 6 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 60 | 63
mmol/L | 4.954 (0.826) | 5.089 (0.731)

14. Post Hoc Outcome: Event Rate of "All Confirmed Low CGMS Excursions" (Individual Component of Primary Endpoint) Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years (Events Per Patient-year)
Description: "All confirmed low CGMS excursions" consisted of all low continuous glucose monitoring system (CGMS) excursions (interstitial glucose <70 mg/dL [3.9 mmol/L]) confirmed by fingerstick blood glucose (FSBG) <70 mg/dL.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
events per patient-year | 74.61 (74.09) | 71.60 (53.20)

15. Post Hoc Outcome: Event Rate of "All Confirmed Low FSBG" (Individual Component of the Primary Endpoint) Defined as the Total Number of Episodes Divided by the Total Duration of the On-treatment Period in Years (Events Per Patient-year)
Description: "All confirmed low FSBG" consisted of all low FSBG readings (values <70 mg/dL) performed at other times.
Time Frame: 6 months
Population: Same as for primary endpoint: mITT population.
Measure: Mean (Standard Deviation); unit: events per patient-year
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 61 | 64
events per patient-year | 192.69 (121.78) | 168.24 (101.21)

16. Other Pre Specified Outcome: Nocturnal Blood Glucose Variability Based on All On-treatment CGMS Values
Description: Calculated for any given patient as the standard deviation (SD) of all CGMS interstitial glucose values recorded during the nocturnal time period (between 23:00 and 07:00 hours).
Time Frame: 6 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lantus (Insulin Glargine) | NPH Insulin
Number analyzed (Participants) | 60 | 63
mmol/L | 4.747 (0.973) | 4.837 (0.825)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline to 7 days after last treatment visit.
Description: The safety analyses were conducted according to the treatment received rather than according to the randomization groups.
Arm/Group | Lantus | NPH Insulin
Serious Adverse Events (participants affected / at risk) | 8/62 | 2/63
Other Adverse Events (participants affected / at risk) | 30/62 | 33/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lantus (N=62) | NPH Insulin (N=63)
Viral infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lantus (N=62) | NPH Insulin (N=63)
Gastroenteritis (Infections and infestations) | 6 | 6
Nasopharyngitis (Infections and infestations) | 6 | 5
Pharyngitis (Infections and infestations) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 3 | 5
Otitis media (Infections and infestations) | 1 | 4
Tonsillitis (Infections and infestations) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 5 | 4
Device lead damage (General disorders) | 5 | 2
Pyrexia (General disorders) | 3 | 7

LIMITATIONS AND CAVEATS:
There are numerous potential biases that could affect the timing and frequency of performance of sporadic FSBG, such as mealtime dosing and choice of bolus insulin dose, stability and familiarity with insulin regimens, and parental anxiety levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.